CLINICAL TRIAL: NCT01215643
Title: A Multicenter, Randomized, Open Label, Parallel-group Phase IIB Study on the Efficacy and Safety of Oral Regimens of DEB025 Alone or in Combination With Ribavirin Versus Standard of Care (Peg-IFNα2a Plus Ribavirin) in Treatment-naïve Hepatitis C Genotype 2 and 3 Patients
Brief Title: Efficacy and Safety of Alisporivir Alone or Combined With RBV or PEG in Chronic Hepatitis C Genotype 2 and 3 Treatment-naïve Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDEB025A2211; 2010-020034-26 (EudraCT Number)
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C; Chronic Pain
Keywords: Chronic hepatitis C genotype 2; Chronic hepatitis C genotype 3; Cyclophilin inhibitor
MeSH Terms: conditions — Hepatitis C; Chronic Pain | interventions — alisporivir; peginterferon alfa-2a; Ribavirin

ARMS (5):
- ALV 1000 mg (Experimental): Alisporivir (ALV) 600 mg twice daily (BID) for 1 week, followed by ALV 1000 mg once daily (QD) during Weeks 2 to 24.
  Interventions: Drug: Alisporivir
- ALV 600 mg+RBV (Experimental): Alisporivir (ALV) 600 mg BID with RBV for 1 week, followed by ALV 600 mg QD with ribavirin (RBV) during Weeks 2 to 24.
  Interventions: Drug: Alisporivir; Drug: Ribavirin
- ALV 800 mg+RBV (Experimental): Alisporivir (ALV) 600 mg BID with RBV for 1 week, followed by ALV 800 mg QD with RBV during Weeks 2 to 24.
  Interventions: Drug: Alisporivir; Drug: Ribavirin
- ALV 600 mg+PEG (Experimental): Alisporivir (ALV) 600 mg BID with Peginterferon alfa-2a (PEG) for 1 week, followed by ALV 600 mg QD with PEG once weekly during Weeks 2 to 24.
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a
- PEG+RBV (Active Comparator): Peginterferon alfa-2a (PEG) and RBV during Weeks 1 to 24.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Alisporivir — ALV 200 mg soft gel capsules administered orally
  Other Names: DEB025; ALV
  Arms: ALV 1000 mg; ALV 600 mg+PEG; ALV 600 mg+RBV; ALV 800 mg+RBV
Drug: Peginterferon alfa-2a — PEG 180 μg administered via subcutaneous (s.c.) injection once weekly
  Other Names: Pegasys®; PEG
  Arms: ALV 600 mg+PEG; PEG+RBV
Drug: Ribavirin — RBV 400 mg (2 x 200 mg tablets) administered orally twice daily (BID)
  Other Names: Copegus®; RBV
  Arms: ALV 600 mg+RBV; ALV 800 mg+RBV; PEG+RBV

SUMMARY:
The study is to investigate whether alisporivir (ALV; DEB025) alone or in combination with either ribavirin (RBV) or peginterferon alfa-2a (PEG) is more efficient compared to standard of care (PEG+RBV) in treatment-naïve participants with hepatitis C virus (HCV) genotype 2 and 3. In addition, triple therapy with DEB025 plus standard of care will be applied to participants not achieving rapid viral response (RVR) in the different arms.

ELIGIBILITY:
Inclusion criteria:

* Chronic hepatitis C viral infection
* Plasma HCV RNA level lower limit ≥ 10,000 IU/ml assessed by quantitative polymerase chain reaction (qPCR) or equivalent at screening (no upper limit)
* HCV genotype 2 or 3
* No previous treatment for hepatitis C infection

Exclusion criteria:

* Evidence of cirrhosis at the time of screening
* Evidence of hepatocellular carcinoma at the time of screening
* Any other cause of relevant liver disease other than HCV
* Alanine aminotransferase (ALT) ≥ 10 times upper limit of normal (ULN)
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (69):
- United States (16):
  - Scripps Clinic, La Jolla, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - Research and Education Inc., San Diego, California
  - Island View Gastroenterology Associates, Ventura, California
  - Hawai Medical Center East LLC, Honolulu, Hawaii
  - Cotton O'Neil Clinical Research, Topeka, Kansas
  - The Office of Dr. Claudia Martorell, Springfield, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - The North Texas Research Institute, Arlington, Texas
  - Liver Associates of Texas, Houston, Texas
  - Liver Specialist of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
- Australia (6):
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Center, Greenslopes, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
- France (4):
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
- India (9):
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Guwahati
  - Novartis Investigative Site, Haryāna
  - Novartis Investigative Site, Hyderabad - Andhra Pradesh
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
- Italy (5):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Pavia
  - Novartis Inestigative Site, Roma
  - Novartis Investigative Site, Torino
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lódz
  - Novartis Investigative Site, Warsaw
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- South Korea (4):
  - Novartis Korea Ltd., Seoul, Seoul
  - Novartis Inestigative Center, Pusan
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
- Taiwan (5):
  - Novartis Investigative Site, Douliu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Niaosong Township
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Songkhla
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Plymouth

REFERENCES:
- [Result] Pawlotsky JM, Flisiak R, Sarin SK, Rasenack J, Piratvisuth T, Chuang WL, Peng CY, Foster GR, Shah S, Wedemeyer H, Hezode C, Zhang W, Wong KA, Li B, Avila C, Naoumov NV; VITAL-1 study team. Alisporivir plus ribavirin, interferon free or in combination with pegylated interferon, for hepatitis C virus genotype 2 or 3 infection. Hepatology. 2015 Oct;62(4):1013-23. doi: 10.1002/hep.27960. Epub 2015 Aug 10. PMID 26118427

RESULTS

PARTICIPANT FLOW:
Groups:
- ALV 600 mg+RBV: ALV 600 mg BID with ribavirin (RBV) for 1 week, followed by ALV 600 mg QD with RBV during Weeks 2 to 24.
- ALV 800 mg+RBV: ALV 600 mg BID with RBV for 1 week, followed by ALV 800 mg QD with RBV during Weeks 2 to 24.
- ALV 600 mg+PEG: ALV 600 mg BID with PEG for 1 week, followed by ALV 600 mg QD with peginterferon alfa-2a (PEG) during Weeks 2 to 24.
- PEG+RBV: PEG and RBV during Weeks 1 to 24.
Period: Overall Study
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Started | 83 | 84 | 94 | 39 | 40
Completed | 74 | 80 | 82 | 35 | 29
Not Completed | 9 | 4 | 12 | 4 | 11

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- ALV 1000 mg: ALV 600 mg BID for 1 week, followed by ALV 1000 mg QD during Weeks 2 to 24.
- ALV 600 mg+RBV: ALV 600 mg BID with RBV for 1 week, followed by ALV 600 mg QD with RBV during Weeks 2 to 24.
- ALV 600 mg+PEG: ALV 600 mg BID with PEG for 1 week, followed by ALV 600 mg QD with PEG during Weeks 2 to 24.
- Total: Total of all reporting groups
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV | Total
Number analyzed (Participants) | 83 | 84 | 94 | 39 | 40 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.27) | 42.8 (11.77) | 42.6 (11.00) | 43.2 (10.56) | 39.9 (11.20) | 41.8 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 33 | 14 | 16 | 123
  Male | 51 | 56 | 61 | 25 | 24 | 217

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Rapid Viral Response (RVR) After 4 Weeks of Treatment < the Limit of Quantification (RVR4LOQ)
Description: RVR4LOQ was defined as RVR [serum hepatitis C virus (HCV) ribonucleic acid (RNA) < the limit of quantification (LOQ), i.e., < 25 IU/mL], after 4 weeks of treatment.
Time Frame: after 4 weeks of treatment
Population: Full Analysis Set (FAS), defined as all participants to whom study treatment was correctly assigned.
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants | 28.4 | 36.9 | 41.9 | 84.6 | 72.5

2. Secondary Outcome: Percentage of Participants With RVR After 4 Weeks of Treatment < the Limit of Detection (RVR4LOD)
Description: RVR4LOD was defined as Rapid Viral Response (RVR) [serum HCV RNA < the limit of detection (LOD), i.e., < 10 IU/mL], after 4 weeks of treatment.
Time Frame: after 4 weeks of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants | 18.5 | 14.3 | 23.7 | 69.2 | 60.0

3. Secondary Outcome: Percentage of Participants With RVR4LOQ and RVR4LOD (Genotype 2)
Time Frame: after 4 weeks of treatment
Population: Participants in the Full Analysis Set with genotype 2 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 23 | 30 | 26 | 11 | 13
percentage of participants
  RVR4LOQ | 21.7 | 23.3 | 46.2 | 81.8 | 76.9
  RVR4LOD | 13.0 | 10.0 | 26.9 | 63.6 | 53.8

4. Secondary Outcome: Percentage of Participants With RVR4LOQ and RVR4LOD (Genotype 3)
Time Frame: after 4 weeks of treatment
Population: Participants in the Full Analysis Set with genotype 3 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 58 | 54 | 67 | 28 | 27
percentage of participants
  RVR4LOQ | 31.0 | 44.4 | 40.3 | 85.7 | 70.4
  RVR4LOD | 20.7 | 16.7 | 22.4 | 71.4 | 63.0

5. Secondary Outcome: Percentage of Participants With Complete Early Viral Response (cEVR) After 12 Weeks of Treatment (cEVR12LOQ and cEVR12LOD)
Description: cEVR12LOQ and cEVR12LOD were defined as cEVR [serum HCV RNA < LOQ and < LOD] after 12 weeks of treatment, respectively.
Time Frame: after 12 weeks of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants
  cEVR12LOQ | 93.8 | 95.2 | 90.3 | 94.9 | 85.0
  cEVR12LOD | 91.4 | 86.9 | 90.3 | 84.6 | 82.5

6. Secondary Outcome: Percentage of Participants With cEVR12LOQ and cEVR12LOD (Genotype 2)
Time Frame: after 12 weeks of treatment
Population: Participants in the Full Analysis Set with genotype 2 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 23 | 30 | 26 | 11 | 13
percentage of participants
  cEVR12LOQ | 100.0 | 96.7 | 80.8 | 100.0 | 84.6
  cEVR12LOD | 100.0 | 83.3 | 80.8 | 90.9 | 84.6

7. Secondary Outcome: Percentage of Participants With cEVR12LOQ and cEVR12LOD (Genotype 3)
Time Frame: after 12 weeks of treatment
Population: Participants in the Full Analysis Set with genotype 3 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 58 | 54 | 67 | 28 | 27
percentage of participants
  cEVR12LOQ | 91.4 | 94.4 | 94.0 | 92.9 | 85.2
  cEVR12LOD | 87.9 | 88.9 | 94.0 | 82.1 | 81.5

8. Secondary Outcome: Percentage of Participants With End of Treatment Response (ETR) Within 24 Weeks (ETR24LOQ and ETR24LOD)
Description: ETR24LOQ and ETR24LOD were defined as ETR [serum HCV RNA < LOQ and < LOD] after 24 weeks of treatment or when prematurely discontinued.
Time Frame: at end of treatment, within 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants
  ETR24LOQ | 95.1 | 96.4 | 95.7 | 94.9 | 87.5
  ETR24LOD | 92.6 | 94.0 | 92.5 | 92.3 | 82.5

9. Secondary Outcome: Percentage of Participants With ETR24LOQ and ETR24LOD (Genotype 2)
Time Frame: at end of treatment, within 24 weeks
Population: Participants in the Full Analysis Set with genotype 2 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 23 | 30 | 26 | 11 | 13
percentage of participants
  ETR24LOQ | 100.0 | 96.7 | 84.6 | 100.0 | 92.3
  ETR24LOD | 100.0 | 96.7 | 76.9 | 100.0 | 84.6

10. Secondary Outcome: Percentage of Participants With ETR24LOQ and ETR24LOD (Genotype 3)
Time Frame: at end of treatment, within 24 weeks
Population: Participants in the Full Analysis Set with genotype 3 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 58 | 54 | 67 | 28 | 27
percentage of participants
  ETR24LOQ | 93.1 | 96.3 | 100.0 | 92.9 | 85.2
  ETR24LOD | 89.7 | 92.6 | 98.5 | 89.3 | 81.5

11. Secondary Outcome: Percentage of Participants With RVR Who Achieved Sustained Viral Response (SVR) 12 Weeks After the End of Treatment (SVR12LOQ and SVR12LOD)
Description: SVR12LOQ and SVR12LOD were defined as Sustained Viral Response (SVR) [serum HCV RNA < LOQ and < LOD] 12 weeks after treatment, respectively.
Time Frame: 12 weeks after the end of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants
  SVR12LOQ | 81.5 | 84.5 | 80.6 | 76.9 | 62.5
  SVR12LOD | 80.2 | 84.5 | 80.6 | 74.4 | 60.0

12. Secondary Outcome: Percentage of Participants With RVR Who Achieved SVR12LOQ and SVR12LOD (Genotype 2)
Time Frame: 12 weeks after the end of treatment
Population: Participants in the Full Analysis Set with genotype 2 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 23 | 30 | 26 | 11 | 13
percentage of participants
  SVR12LOQ | 78.3 | 76.7 | 76.9 | 72.7 | 61.5
  SVR12LOD | 78.3 | 76.7 | 76.9 | 72.7 | 53.8

13. Secondary Outcome: Percentage of Participants With RVR Who Achieved SVR12LOQ and SVR12LOD (Genotype 3)
Time Frame: 12 weeks after the end of treatment
Population: Participants in the Full Analysis Set with genotype 3 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 58 | 54 | 67 | 28 | 27
percentage of participants
  SVR12LOQ | 82.8 | 88.9 | 82.1 | 78.6 | 63.0
  SVR12LOD | 81.0 | 88.9 | 82.1 | 75.0 | 63.0

14. Secondary Outcome: Percentage of Participants With RVR Who Achieved SVR at 24 Weeks After the End of Treatment (SVR24LOQ and SVR24LOD)
Time Frame: 24 weeks after the end of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants
  SVR24LOQ | 80.2 | 84.5 | 80.6 | 79.5 | 57.5
  SVR24LOD | 80.2 | 84.5 | 79.6 | 79.5 | 57.5

15. Secondary Outcome: Percentage of Participants With RVR Who Achieved SVR24LOQ and SVR24LOD (Genotype 2)
Time Frame: 24 weeks after the end of treatment
Population: Participants in the Full Analysis Set with genotype 2 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 23 | 30 | 26 | 11 | 13
percentage of participants
  SVR24LOQ | 78.3 | 76.7 | 76.9 | 72.7 | 53.8
  SVR24LOD | 78.3 | 76.7 | 76.9 | 72.7 | 53.8

16. Secondary Outcome: Percentage of Participants With RVR Who Achieved SVR24LOQ and SVR24LOD (Genotype 3)
Time Frame: 24 weeks after the end of treatment
Population: Participants in the Full Analysis Set with genotype 3 HCV infection
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 58 | 54 | 67 | 28 | 27
percentage of participants
  SVR24LOQ | 81.0 | 88.9 | 82.1 | 82.1 | 59.3
  SVR24LOD | 81.0 | 88.9 | 80.6 | 82.1 | 59.3

17. Secondary Outcome: Percentage of Participants With On-treatment Viral Breakthrough
Description: Viral breakthrough was defined as either:
  * Confirmed increase of HCV RNA ≥1 log10 above nadir (nadir = lowest HCV RNA value during treatment), or
  * HCV RNA becoming ≥ 100 IU/mL after previously being undetectable (< LOD) during treatment
Time Frame: within 24 weeks of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants | 2.5 | 3.6 | 2.2 | 5.1 | 0.0

18. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as having reappearance of detectable HCV RNA after previously being undetectable (< LOD) during treatment.
Time Frame: within 24 weeks after the end of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ALV 1000 mg | ALV 600 mg+RBV | ALV 800 mg+RBV | ALV 600 mg+PEG | PEG+RBV
Number analyzed (Participants) | 81 | 84 | 93 | 39 | 40
percentage of participants
  0 to 12 weeks after the end of treatment | 9.9 | 8.3 | 6.5 | 10.3 | 20.0
  12 to 24 weeks after the end of treatment | 1.2 | 0.0 | 0.0 | 0.0 | 5.0

ADVERSE EVENTS:
Groups:
- ALV 1000 mg: On-treatment AEs: Adverse events (AEs) occurring while on treatment in participants receiving ALV 600 mg BID for 1 week, followed by ALV 1000 mg QD during Weeks 2 to 24.
- ALV 600 mg+RBV: On-treatment AEs: AEs occurring while on treatment in participants receiving ALV 600 mg BID with RBV for 1 week, followed by ALV 600 mg QD with RBV during Weeks 2 to 24.
- ALV 800 mg+RBV: On-treatment AEs: AEs occurring while on treatment in participants receiving ALV 600 mg BID with RBV for 1 week, followed by ALV 800 mg QD with RBV during Weeks 2 to 24.
- ALV 600 mg+PEG: On-treatment AEs: AEs occurring while on treatment in participants receiving ALV 600 mg BID with PEG for 1 week, followed by ALV 600 mg QD with PEG during Weeks 2 to 24.
- PEG+RBV: On-treatment AEs: AEs occurring while on treatment in participants receiving PEG and RBV during Weeks 1 to 24.
- ALV 1000 mg: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 600 mg BID for 1 week, followed by ALV 1000 mg QD during Weeks 2 to 24.
- ALV 600 mg+RBV: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 600 mg BID with RBV for 1 week, followed by ALV 600 mg QD with RBV during Weeks 2 to 24.
- ALV 800 mg+RBV: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 600 mg BID with RBV for 1 week, followed by ALV 800 mg QD with RBV during Weeks 2 to 24.
- ALV 600 mg+PEG: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 600 mg BID with PEG for 1 week, followed by ALV 600 mg QD with PEG during Weeks 2 to 24.
- PEG+RBV: Post-treatment AEs: AEs occurring after end of treatment in participants receiving PEG and RBV during Weeks 1 to 24.
Arm/Group | ALV 1000 mg: On-treatment AEs | ALV 600 mg+RBV: On-treatment AEs | ALV 800 mg+RBV: On-treatment AEs | ALV 600 mg+PEG: On-treatment AEs | PEG+RBV: On-treatment AEs | ALV 1000 mg: Post-treatment AEs | ALV 600 mg+RBV: Post-treatment AEs | ALV 800 mg+RBV: Post-treatment AEs | ALV 600 mg+PEG: Post-treatment AEs | PEG+RBV: Post-treatment AEs
Serious Adverse Events (participants affected / at risk) | 4/82 | 1/84 | 9/94 | 4/39 | 2/37 | 2/82 | 4/84 | 1/94 | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 64/82 | 69/84 | 76/94 | 37/39 | 30/37 | 10/82 | 10/84 | 13/94 | 5/39 | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALV 1000 mg: On-treatment AEs (N=82) | ALV 600 mg+RBV: On-treatment AEs (N=84) | ALV 800 mg+RBV: On-treatment AEs (N=94) | ALV 600 mg+PEG: On-treatment AEs (N=39) | PEG+RBV: On-treatment AEs (N=37) | ALV 1000 mg: Post-treatment AEs (N=82) | ALV 600 mg+RBV: Post-treatment AEs (N=84) | ALV 800 mg+RBV: Post-treatment AEs (N=94) | ALV 600 mg+PEG: Post-treatment AEs (N=39) | PEG+RBV: Post-treatment AEs (N=37)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALV 1000 mg: On-treatment AEs (N=82) | ALV 600 mg+RBV: On-treatment AEs (N=84) | ALV 800 mg+RBV: On-treatment AEs (N=94) | ALV 600 mg+PEG: On-treatment AEs (N=39) | PEG+RBV: On-treatment AEs (N=37) | ALV 1000 mg: Post-treatment AEs (N=82) | ALV 600 mg+RBV: Post-treatment AEs (N=84) | ALV 800 mg+RBV: Post-treatment AEs (N=94) | ALV 600 mg+PEG: Post-treatment AEs (N=39) | PEG+RBV: Post-treatment AEs (N=37)
Anaemia (Blood and lymphatic system disorders) | 8 | 11 | 10 | 4 | 3 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 2 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 8 | 13 | 10 | 4 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 3 | 6 | 2 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 6 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1 | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 5 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 4 | 7 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6 | 7 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 8 | 3 | 0 | 2 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 6 | 10 | 9 | 1 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 8 | 7 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 5 | 0 | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 17 | 15 | 23 | 9 | 5 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 7 | 7 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 10 | 7 | 11 | 3 | 8 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 5 | 3 | 5 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 21 | 23 | 30 | 18 | 10 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 8 | 6 | 9 | 8 | 4 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 2 | 5 | 8 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 2 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 3 | 3 | 5 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 14 | 16 | 15 | 12 | 9 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 2 | 5 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 5 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 4 | 4 | 3 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 4 | 2 | 4 | 3 | 4 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 14 | 14 | 10 | 9 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 15 | 10 | 5 | 2 | 3 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 10 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3 | 2 | 1 | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 7 | 13 | 8 | 8 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 3 | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 11 | 16 | 5 | 4 | 1 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 19 | 18 | 27 | 16 | 7 | 0 | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 3 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 8 | 9 | 5 | 1 | 5 | 1 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 2 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 12 | 7 | 9 | 3 | 3 | 0 | 0 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 12 | 14 | 4 | 6 | 0 | 2 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 4 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 13 | 12 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 8 | 4 | 9 | 7 | 0 | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 5 | 6 | 3 | 3 | 1 | 1 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 14 | 12 | 7 | 6 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 9 | 14 | 2 | 3 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 9 | 10 | 8 | 5 | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other